CLINICAL TRIAL: NCT00378261
Title: A Multicenter, Randomized, Open Study to Evaluate the Impact of an Electronic Data Capture System on the Care of Patients With Rheumatoid Arthritis
Brief Title: APART Advanced Profiling of Anti-Rheumatic Therapies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centocor Ortho Biotech Services, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CR004807
Record Dates: First submitted 2006-09-15; First posted 2006-09-19 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-04

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Treatment Outcome

INTERVENTIONS:
Procedure: Use of an Electronic Data Capture System by patients and physicians to assess patient-physician interactions & therapeutic decisions & outcomes in RA subjects.

SUMMARY:
The purpose of this study is to evaluate the utility of an electronic data capture system (EDCS) in a rheumatology clinical practice setting and to assess the impact of this system on patient satisfaction with patient-physician interaction.

DETAILED DESCRIPTION:
This is a randomized, multicenter observational study to assess the impact of the EDCS in a rheumatology clinical practice setting on patient satisfaction with patient-physician communication using the Health Tracker electronic data capture system . Patients will be randomly assigned in a 2:1 ratio to the Health Tracker-user or non-user groups, respectively. The primary outcomes of this study will be the impact that information gathered and analyzed by an electronic data capture system has on patient satisfaction with arthritis care and patient physician interactions in clinical practice. Patient satisfaction will be assessed using a questionnaire developed specifically for this study.

This study does not involve the use of any investigational drugs, and the protocol does not mandate the treatment regimen patients will receive. Physicians will prescribe antirheumatic medications in accordance with usual clinical practice. The planned duration of subject participation is 12 months

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with active rheumatoid arthritis according to the revised criteria of the ACR (1987)
* Have rheumatoid arthritis that requires regularly scheduled visits with their rheumatologist at least every 3 months
* Willing and able to adhere to protocol requirements and participate in a study, lasting 12 months

Exclusion Criteria:

* Patients currently receiving investigational drugs
* Currently participating in other clinical trials or safety registries for rheumatoid arthritis or rheumatoid arthritis -related therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1079 (Actual)
Dates: Start 2004-01; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Primary endpoints for the Health Tracker-user group are the change in the patient satisfaction and patient-physician interaction surveys between the pre- and post-randomization phases.

SECONDARY OUTCOMES:
Changes between the pre- and post-randomization phases in the following clinical evaluations: HAQ scores, SF-12 scores, Patient assessed painful and/or swollen joint counts, Health care professional assessed tender and swollen joint counts

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.

REFERENCES:
- See also: A Multicenter, Randomized, Open Study to Evaluate the Impact of an Electronic Data Capture System on the Care of Patients with Rheumatoid Arthritis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=130&filename=CR004807_CSR.pdf